CLINICAL TRIAL: NCT06882681
Title: Novel Micellar Formulation of Silymarin with Enhanced Bioavailability in a Double-Blind, Randomized, Crossover Human Trial
Brief Title: Silymarin Bioavailability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-11-002S
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Bioavailability and Pharmacokinetics
Keywords: milk thistle; silymarin; LipoMicel; pharmacokinetics; bioavailability; absorption; micelles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LipoMicel Milk Thistle (Experimental): Participants receive their treatment of a novel micellar Milk Thistle formulation (i.e, LipoMicel soft-gel capsules) at a total dose of approx. 140 mg of silymarins per capsule. Treatments are consumed with a glass of water (approx. 125mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of 1 week between each treatment is used.
  Interventions: Dietary Supplement: LipoMicel Milk Thistle
- Unformulated/Standard Milk Thistle Extract (Experimental): Participants receive their treatment of standard/unformulated Milk Thistle (i.e, hard-gel capsules) at a total dose of approx. 130 mg of silymarins per capsule. Treatments are consumed with a glass of water (approx. 125mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of 1 week between each treatment is used.
  Interventions: Dietary Supplement: Unformulated Milk Thistle Extract

INTERVENTIONS:
Dietary Supplement: LipoMicel Milk Thistle — A maximum single dose of approx. 140 mg silymarin (in soft gel capsule)
  Arms: LipoMicel Milk Thistle
Dietary Supplement: Unformulated Milk Thistle Extract — A maximum single dose of approx. 130 mg silymarin (in hard gel capsules)
  Arms: Unformulated/Standard Milk Thistle Extract

SUMMARY:
This study seeks to evaluate and compare the pharmacokinetics of a novel micellar silymarin formulation with that of a standard silymarin formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 21- 65 years
* Healthy, good physical condition
* Voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Serious acute or chronic diseases e.g. liver, kidney, or gastrointestinal diseases
* Contraindication or allergies to milk thistle
* Pregnancy or breastfeeding
* Concurrent use of supplements and/or medications
* Participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested silymarin in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of other capsules containing silymarin.
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested silymarin in healthy adult volunteers and compare the peak plasma concentration (Cmax) with that of other capsules containing silymarin.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested silymarin in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax) with that of other capsules containing silymarin.
MRT: Mean residence time | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested silymarin in healthy adult volunteers and compare the mean residence time (MRT) with that of other capsules containing silymarin.
T1/2: elimination half-life | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested silymarin in healthy adult volunteers and compare the elimination half-life (T1/2) with that of other capsules containing silymarin.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, PhD, Principal Investigator — Isura
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No